CLINICAL TRIAL: NCT04184206
Title: Effects of Attention Training Interventions on Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Moved institutions, study terminated
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Matthew Sacchet, Assistant Neuroscientist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: McLean
Record Dates: First submitted 2019-04-04; First posted 2019-12-03 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Depression; Attention Training; Symptoms, Cognitive; Symptoms, Affective; Symptoms, Behavioral
MeSH Terms: conditions — Depression; Neurobehavioral Manifestations; Affective Symptoms; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- attention training intervention 1 (Active Comparator): 14-day smartphone-based audio-guided attention training program with heavy mindfulness influence
  Interventions: Behavioral: attention training intervention 1
- attention training intervention 2 (Active Comparator): 14-day smartphone-based audio-guided attention training program with moderate mindfulness influence
  Interventions: Behavioral: attention training intervention 2
- attention training intervention 3 (Active Comparator): 14-day smartphone-based audio-guided intervention without mindfulness emphasis
  Interventions: Behavioral: attention training intervention 3

INTERVENTIONS:
Behavioral: attention training intervention 1 — 14-day smartphone-based audio-guided attention training program with heavy mindfulness component
  Arms: attention training intervention 1
Behavioral: attention training intervention 2 — 14-day smartphone-based audio-guided attention training program with moderate mindfulness component
  Arms: attention training intervention 2
Behavioral: attention training intervention 3 — 14-day smartphone-based audio-guided attention training program without mindfulness component
  Arms: attention training intervention 3

SUMMARY:
The purpose of this study is to study the effects of attention training interventions on symptoms and brain function in major depressive disorder.

DETAILED DESCRIPTION:
Attention training programs including mindfulness meditation-based interventions have been shown to be effective for treating depression. Currently the biological and psychological mechanisms of action of attention training for major depression disorder are unknown. The objective of the current study is to improve the investigator's understanding of the mechanisms of attention training interventions for depression.

Research participants will include approximately 165 individuals with major depressive disorder randomized to one of three types of attention training programs. Before and after intervention participants will complete a number of biological assessments including MRI, EEG, behavioral tasks, and questionnaires. The study will be completed across three visits: (1) a screening visit; (2) data collection session 1; and (3) data collection session 2.

ELIGIBILITY:
Inclusion Criteria include:

* DSM-5 criteria for major depressive disorder
* Written informed consent
* Both biological sexes, any ethnicity
* Age 18-55
* Scores exceeding cutoffs on depression questionnaires
* Right-handed
* Normal or corrected-to-normal vision and hearing
* Fluency in written and spoken English
* Absence of psychotropic medication

Exclusion Criteria include:

* Use of substances or prior treatments that may interfere with study procedures or outcomes (e.g., stimulants, blood pressure medication)
* Medical conditions that may interfere with study procedures or outcomes (e.g., thyroid disorder)
* Current therapy and practices overlapping with study interventions
* Select other DSM-5 disorders and symptoms (e.g., psychotic symptoms, suicidal ideation)
* Failure to meet MRI safety requirements or suitability
* Significant inconsistencies in self-report or first-degree relatives with history or current psychotic symptoms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
changes in questionnaire measures including severity of depression (e.g., Beck Depression Inventory [BDI-II]: minimum/maximum values = 0/63, higher scores indicate worse outcome) | pre-treatment to post-treatment (approximately 3-4 weeks from intervention start date)
changes in neural measures including "functional connectivity" functional magnetic resonance imaging (fMRI) collected during rest conditions | pre-treatment to post-treatment (approximately 3-4 weeks from intervention start date)
changes in behavioral task performance including related to affective (e.g., Probabilistic Reward Task [PRT]) | pre-treatment to post-treatment (approximately 3-4 weeks from intervention start date)
changes in behavioral task performance including related to cognitive processing (e.g., Flanker Task). | pre-treatment to post-treatment (approximately 3-4 weeks from intervention start date)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No